CLINICAL TRIAL: NCT06759402
Title: Family-based Telemedicine vs. Inpatient Anorexia Nervosa Treatment (FIAT)
Acronym: FIAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bielefeld University (Other); Techniker Krankenkasse (Other); BARMER (Other); AOK Niedersachsen (Unknown); Mobil Krankenkasse (Unknown); Meine Krankenkasse (Unknown); Medicalnetworks CJ GmbH & Co.KG (Unknown); AOK Baden-Württemberg (Industry); DAK Gesundheit (Other); BIG-direkt (Unknown); mhplus (Unknown); Bahn-BKK (Unknown); OFFIS - Institut für Informatik (Unknown); Prof. Daniel Le Grange, UCSF (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med Christoph Correll, Clinic Director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2/114/24
Record Dates: First submitted 2024-12-09; First posted 2025-01-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Anorexia Nervosa; Anorexia in Adolescence
Keywords: Psychotherapy; Family Based Treatment; RCT; Inpatient Treatment
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: multicentred, longitudinal, randomized controlled non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FBT (Experimental): family-based therapy as a stepped care model using telemedicine
  Interventions: Behavioral: Family based treatment
- IMT (Active Comparator): inpatient multimodal therapy
  Interventions: Behavioral: Inpatient multimodal therapy

INTERVENTIONS:
Behavioral: Family based treatment — FBT is an intensive, manualized therapy in which the parents of those affected are closely involved in a resource-oriented manner by FBT-certified therapists. FBT takes place in 3 phases: in phase 1, the parents take responsibility for their child's weight gain. Phase 2 involves the gradual transfer of responsibility for eating back to the patient. Phase 3 focuses on individual issues of the children and adolescents, e.g. catching up on important developmental steps missed due to the illness.
  Arms: FBT
Behavioral: Inpatient multimodal therapy — comprehensive, patient-oriented and multidisciplinary approach to address eating disorders following the S3 joint German treatment guidelines in specialized hospitals. Includes individual psychotherapy, family sessions, body-oriented therapy, nutritional counseling, group therapy sessions, relaxation techniques, mindfulness practices, and skills training. Targeted weight gain per week is at least 500g.
  Arms: IMT

SUMMARY:
The FIAT study is funded by the Innovationsfonds of the German Ministry of Health via the DLR Project Management Agency. The study will be conducted in up to 21 hospitals across Germany and in collaboration with 10 German public health insurance companies. The primary aim of this study is to compare Family-Based Treatment delivered via telehealth (FBT) with inpatient multimodal therapy (IMT) with respect to treatment outcomes and health economic data. The results of the study will serve as a basis for the decision on the inclusion of FBT in the German S3 guidelines and the future reimbursement of FBT by public health insurances in Germany.

ELIGIBILITY:
Inclusion Criteria:

* restrictive and bulimic subtypes of anorexia nervosa (ICD-10: F50.00; F50.01)
* inpatient treatment indication according to S3 guideline
* weight < 3. BMI-percentile or
* weight <10. percentile and psychiatric comorbidity/rapid weight loss/lack of weight gain during outpatient treatment over last three month
* planned inpatient treatment
* insured with one of the participating health insurance companies
* stable internet connection

Exclusion Criteria:

* weight <67%mBMI
* acute self harm or danger to others
* acute psychosis or suicidal tendencies
* current substance abuse
* child abuse or domestic violence in the family
* insured with other health insurance company
* judicial placement order for inpatient treatment
* known, currently existing child protection problems or proceedings by the family court

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in %mBMI | 12 months
  The %mBMI is calcualted based on bodyweight and height, measured by the study team. Change is the difference between the baseline and 12 month %mBMI.

SECONDARY OUTCOMES:
Specific psychopathology for anorexia nervosa | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the eating disorder examination-questionnaire (EDE-Q). The scores of the EDE-Q are presented on a scale between 0 and 6, where higher scores mean higher presence of symptoms.
Compulsive exercise | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the compulsive exercise test (CET). Items are rated on a 6-point Likert type scale from 0 (never true) to 5 (always true), with higher scores correspond with stronger symptoms.
Depression | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the Revised Children's Anxiety and Depression Scale (RCADS). Scores are presented between 0 (never) to 3 (always). The total score is converted into a T-score. Higher T-scores indicate higher presence of symptoms.
Occurrence of adverse events | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the modified over aggression scale (MOAS) in addition with a set serious adverse events list. Higher scores on the MOAS indicate more severe cases of aggressive behaviors.
Menstrual status | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by structural interview.
Medication | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by structural interview.
Motivation for change | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the anorexia nervosa stages of change questionnaire (ANSOCQ). Each item can scored between 1 and 5. Higher scores indicate higher levels of motivation.
Insight into illness | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  One item "On a scale of 1 to 10, how severe would you rate yourself as suffering from anorexia?" where a higher score indicates more insight into the illness.
Change in eating disorder quality of life | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the eating disorder quality of life (EDQOL). Each item can be scored on a 6-point scale ranging from 0 ("never") to 5 ("always"). Higher scores indicate lower quality of life.
Change in quality of life | 6 months after baseline and 12 months after baseline.
  Measured by the EQ-5D-Y-5L. Items are scored on 5 levels ("no problems" to "extreme problems") except one, which is scored on a vertical visual analogue scale (endpoints are "the best health you can imagine" and "the worst health you can imagine"). Higher scores indicate more problems.
Emotional and financial burden on the legal guardians | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by the caregiver strain questionnaire (CGSQ-SF11). Items are scored on a 5-point Likert scale (0= not at all, 4= very much). Higher scores indicate greater strain.
Financial burden on the legal guardians | 6 months after baseline and 12 months after baseline.
  Measured by a structured questionnaire about financial strain during treatment. The first question ("Has your child's treatment put a financial strain on you?") is scored on a 4-point Likert scale (1= not at all; 4= extremely). A higher score indicates greater financial strain. The second question ("Have you had any loss of earnings due to your child's illness?") is binary scored (yes/no) and follows up the "yes" condition with the question "how many days were you not able to work?".
Utilization and costs of healthcare services | 6 months after baseline and 12 months after baseline.
  Measured by the Client Service Receipt Inventory (CSRI). Assessing the use of various services in the respective units (e.g., days or hours).
Satisfaction with treatment for patients | At the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months)
  Measured by an adapted version of the treatment satisfaction questionnaire by Lindstedt et al. (2020). The following topics are assessed and scored:
  1. Helpfulness of therapy-elements. Higher scores indicate less helpfulness
  2. Patient-therapist-interaction. Higher scores indicate less positive experiences of interaction.
  3. Treatment goals importance. Higher scores indicate less importance of proposed treatment goals.
  4. Achievement of treatment goals. Higher scores indicate less achievement of proposed treatment goals.
  5. Change in symptoms (before treatment vs. after treatment). Higher scores indicate more positive change in symptoms.
Satisfaction with treatment for parents (Likert scale items) | At the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months)
  Measured by an adapted version of the treatment satisfactory questionnaire by Krautter & Lock (2004). The questions assess the subjective effectiveness of the treatment and treatment satisfaction. Items are scored on all topics on a 5-point Likert scale (0= very ineffective; 4= very effective). Higher scores indicate higher effectiveness. Additionally, the following questions are scored on a 5-point Likert scale (0= not at all; 4= yes, totally) :
  1. "Do you agree that the team that treated your child is competent?"
  2. "Would you recommend this treatment?"
Satisfaction with treatment for parents (Free-text items) | At the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months)
  Measured by an adapted version of the treatment satisfactory questionnaire by Krautter & Lock (2004). The questions assess the subjective effectiveness of the treatment and treatment satisfaction. Two open questions ("What did you find helpful in this treatment?"; "What did you not find helpful in this treatment?") can be answered via free-text.
Suicidality | At the beginning of the study, at the end of treatment (FBT Arm-average: 10 Months; IMT Arm-average: 4 Months; both up to 12 months), 6 months after baseline and 12 months after baseline.
  Measured by asking first whether any suicidal thoughts or behaviors were present in the past 28 days (yes/no). The yes condition is followed up by several questions assessing the presence (yes/no) of:
  * passive suicidal thoughts.
  * active suicidal thoughts.
  * active suicidal thoughts with plan.
  * active suicidal thoughts with plan and preparation.
  * active suicidal thoughts with plan and intention to act upon it.
  * suicidal behaviors, stopped by oneself.
  * suicidal behaviors, stopped by others.
  * suicidal behaviors, carried out, light physical damage.
  * suicidal behaviors, carried out, medium physical damage.
  * suicidal behaviors, carried out, severe physical damage.
  * suicidal behaviors, carried out, death.
  Both children and parents are asked. The children answer for their own thoughts/behaviors, the parents for their child's thoughts/behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Correll, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité- Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krautter, Tonja, and James Lock. "Is manualized family-based treatment for adolescent anorexia nervosa acceptable to patients? Patient satisfaction at the end of treatment." Journal of Family Therapy 26.1 (2004): 66-82.
- [Background] Lindstedt K, Forss E, Elwin M, Kjellin L, Gustafsson SA. Adolescents with full or subthreshold anorexia nervosa in a naturalistic sample: treatment interventions and patient satisfaction. Child Adolesc Psychiatry Ment Health. 2020 May 2;14:16. doi: 10.1186/s13034-020-00323-9. eCollection 2020. PMID 32391079
- [Background] Haas V, Wechsung K, Kaiser V, Schmidt J, Raile K, Busjahn A, Le Grange D, Correll CU. Comparing family-based treatment with inpatient treatment in youth with anorexia nervosa eligible for hospitalization: A 12-month feasibility study. Int J Eat Disord. 2024 Feb;57(2):388-399. doi: 10.1002/eat.24098. Epub 2023 Dec 11. PMID 38082440